CLINICAL TRIAL: NCT01282151
Title: A Randomized Phase III Study of TaxoteRe Plus Cisplatin Versus AlImta Plus Cisplatin in 1st Line Non-squamous Cell Type Lung Cancer
Brief Title: TaxoteRe Plus Cisplatin Versus AlImta Plus Cisplatin in 1st Line Non-squamous Cell Type Lung Cancer
Acronym: TRAIL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruitment due to approval of maintenance pemetrexed treatment
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_05478
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: NSCLC; Non Squamous cell; Docetaxel; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taxotere (Experimental): Docetaxel plus Cisplatin
  Interventions: Drug: Taxotere
- Pemetrexed (Active Comparator): Pemetrexed plus Cisplatin
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Taxotere — Docetaxel 60 mg/m2 q3 weeks Cisplatin 70 mg/m2 q3 weeks
  Other Names: Taxotere(R); Cisplatin
  Arms: Taxotere
Drug: Pemetrexed — Pemetrexed 500 mg/m2 q3 weeks Cisplatin 70 mg/m2 q3 weeks
  Other Names: Alimta (R); Cisplatin
  Arms: Pemetrexed

SUMMARY:
This study is:

* A multicenter, prospective, randomized, phase 3 trial.
* To prove non-inferiority of Taxotere/Cisplatin compared to Pemetrexed/Cisplatin as a front line treatment of patients with non-squamous cell lung cancer.
* 276 patients will be recruited.

DETAILED DESCRIPTION:
Docetaxel is being used in 60mg/m2 3 weekly dosage in Japan and several east Asian institutions. Docetaxel 60mg/m2 and Cisplatin 70 mg/m3 3 weekly regimen will be compared to Pemetrexed 500mg/m2 and Cisplatin 70 mg/m2 3 weekly regimen in first line NSCLC with non-squamous histology.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* ECOG performance status 0-2
* Non-squamous cell type non-small cell lung cancer (NSCLC)
* Stage IV, Stage IIIB cannot be treated with curative intent or Relapsed after surgery or radiation therapy
* No prior chemotherapy except adjuvant chemotherapy and concurrent chemoradiation treatment. The last dose of adjuvant chemotherapy should be at least 6 months earlier from randomization, and the regimen should not contain docetaxel or pemetrexed.
* No prior immunotherapy, biologic therapy
* Measurable lesion with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Hemoglobin >=9.0g/dl, Platelet >=100,000/uL, neutrophil >=1,500 /uL Creatinine <=1.5 x upper normal limit or creatinine clearance >=60 mL/min Bilirubin <=1.5 x upper normal limit, Transaminases <=2 x upper normal limit Alkaline phosphatase <=2 x upper normal limit
* Written informed consent

Exclusion Criteria:

* Pregnancy, Lactating woman
* Woman in child bearing age who refuses to do pregnancy test
* Moderate or greater than grade 1 motor or sensory neurotoxicity
* Hypersensitivity to taxane
* Comorbidity or poor medical conditions
* Other malignancy (except cured basal cell carcinoma or uterine cervical carcinoma in situ)
* Concurrent treatment with other investigational drugs within 30 days before randomization
* Active treatment with other anticancer chemotherapy
* EGFR mutation (exon 19 deletion, L858R, L861Q, G719A/C/S)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | one year
  months after beginning of first cycle chemotherapy

SECONDARY OUTCOMES:
Overall Survival (months from the beginning of first cycle chemotherapy) | three years
  months from the beginning of first cycle chemotherapy
Safety Profile | four months
  Toxicity using CTCAE version 4.0
Response rate | 6-7th week
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Study Chair — Chonnam National University Hospital
Locations (15):
- South Korea (15):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Kyungpook National University Medical Center, Daegu, Kyungpook
  - Hallym University Medical Center, Anyang
  - Dankook University Hospital, Cheonan
  - Keimyung University Dongsan Center, Daegu
  - Yeungnam Univeristy Hospital, Daegu
  - Chosun University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - Inha University Hospital, Incheon
  - Pusan National University Hospital, Pusan
  - Kosin University Gospel Hospital, Pusan
  - Konkuk university medical center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Korea University Medical Center, Seoul
  - Wonju Christian Hospital, Wŏnju